CLINICAL TRIAL: NCT05939102
Title: Eighteen-month Orthodontic Bracket Survival Rate With the Conventional Bonding Technique Versus RMGIC and V-prep: A Split-mouth RCT
Brief Title: Eighteen-month Orthodontic Bracket Survival Rate With the Conventional Bonding Technique Versus RMGIC and V-prep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USJ-2020-010
Record Dates: First submitted 2023-06-30; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Dental Malocclusion
Keywords: resin-modified glass ionomer; surface preparation; orthodontic bracket
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional bracket bonding technique (Active Comparator)
  Interventions: Combination Product: Conventional bracket bonding technique
- V-prep combined with RMGIC for bracket bonding (Experimental)
  Interventions: Combination Product: v-prep combined with RMGIC for bracket bonding

INTERVENTIONS:
Combination Product: v-prep combined with RMGIC for bracket bonding — prepare the tooth surface with the V-prep, then bond a bracket with the RMGIC
  Arms: V-prep combined with RMGIC for bracket bonding
Combination Product: Conventional bracket bonding technique — prepare the tooth with acid-etch, then bond a bracket using resin composite
  Arms: Conventional bracket bonding technique

SUMMARY:
The aim of this study was to evaluate over eighteen months the clinical bonding failure and survival rates of the conventional bonding technique using the Transbond XT (3M Unitek, Monrovia, California, USA) and the RMGIC Fuji Ortho LC (GC Corporation, Tokyo, Japan) prepared with the V-prep. Therefore, one operator using the straight-wire technique bonded two hundred metallic brackets to upper and lower premolars of twenty-five patients requiring an orthodontic treatment. The randomized trial was a single-blind design in a split-mouth comparison. Each patient was randomly allocated one of the two bonding systems for each premolar on each side of the mouth. The bonding and rebonding techniques were standardized throughout the trial and bond failure was recorded each month for a period of eighteen months.

ELIGIBILITY:
Inclusion Criteria:

* require full orthodontic treatment of both arches
* mild or average overbite and crowding
* no restorations on the buccal surface of the premolars

Exclusion Criteria:

* Patients with required extractions in the treatment plan or with poor oral hygiene

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Bracket bonding survival rate | 18 months
  reports of bracket debonding using one of the two bonding techniques

CONTACTS AND LOCATIONS:
Overall Officials: Victor Ghoubril, Ms, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint Joseph University, Beirut, Lebanon

REFERENCES:
- [Background] Ghoubril V, Changotade S, Lutomski D, Ghoubril J, Chakar C, Abboud M, Hardan L, Kharouf N, Khoury E. Cytotoxicity of V-Prep Versus Phosphoric Acid Etchant on Oral Gingival Fibroblasts. J Funct Biomater. 2022 Nov 28;13(4):266. doi: 10.3390/jfb13040266. PMID 36547526
- [Background] Ghoubril V, Ghoubril J, Khoury E. A comparison between RMGIC and composite with acid-etch preparation or hypochlorite on the adhesion of a premolar metal bracket by testing SBS and ARI: In vitro study. Int Orthod. 2020 Mar;18(1):127-136. doi: 10.1016/j.ortho.2019.07.003. Epub 2019 Sep 5. PMID 31495756